CLINICAL TRIAL: NCT00394810
Title: Phase 2 Efficacy and Pharmacodynamic Study of 2-Methoxyestradiol Nanocrystal Colloidal Dispersion(Panzem® NCD) in Patients With Taxane-Refractory, Metastatic,Hormone-Refractory Prostate Cancer
Brief Title: Efficacy and Pharmacodynamic Study of Panzem® NCD in Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-006
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Panzem® NCD

INTERVENTIONS:
Drug: Panzem® NCD — suspension, 100 mg/mL, four times daily continuous dosing

SUMMARY:
This open-label, multicenter, Phase 2 trial, will assess the anti tumor activity, safety and pharmacokinetics, of Panzem® NCD in patients with metastatic, docetaxel refractory, androgen-independent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (pts) must have histologically or cytologically confirmed adenocarcinoma of the prostate.
2. Pts must have evidence of progressive metastatic disease (e.g., new lesions on bone scan or new/enlarging lesions on computerized tomography [CT] scan) or known metastatic disease and rising PSA, during or after treatment with a taxane-based regimen (as well as any other subsequent non-cytotoxic therapy).

   * Pts with bone metastases only (i.e., lacking soft-tissue disease) must have a PSA level of 10 ng/mL or higher.
   * Pts with soft tissue metastases and/or visceral disease must have either measurable disease (per RECIST criteria) or a PSA level of 10 ng/mL or higher.
   * For pts with stable metastatic disease and rising PSA: two consecutive rises in PSA measurement are necessary, each separated from the previous by a minimum of two weeks. The most recent PSA value must be obtained within 1 week prior to registration.
   * At least 3 PSA values within 6 months of registration (each separated by at least 2 weeks) using the same clinical laboratory needs to be available for calculation of the PSA pre-treatment slope. Only those values obtained after the last treatment date (see inclusion criteria #5 below) will be acceptable.
3. Pts must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy with evidence of treatment failure.

   * Pts who have not undergone bilateral orchiectomy must continue their luteinizing hormone-releasing hormone (LHRH) agonist therapy (e.g., leuprolide or goserelin) or LHRH antagonist (e.g. abarelix) while receiving protocol therapy.
   * A serum testosterone level of 50 ng/dL or lower is required to confirm castration status within 4 weeks prior to study entry.
4. For pts previously treated with flutamide (Eulixin), Nilutamide (Nilandron), or bicalutamide (Casodex): pts must have discontinued flutamide 4 weeks or more prior to registration with continued evidence of progressive disease. For bicalutamide or nilutamide, pts must have discontinued the drug 6 weeks or more prior to registration with evidence of progressive disease.

   • Disease progression following anti-androgen withdrawal needs to be confirmed by a rising PSA after the required 4-6 week washout period (e.g. PSA level higher than the last PSA obtained while on anti-androgen therapy).
5. Pts must have received only one prior taxane-based regimen for metastatic disease, with evidence of disease progression (inclusion criteria #2) during treatment or within 6 months of treatment discontinuation. Up to one other prior experimental therapy (non-cytotoxic) is permitted. At least 4 weeks or more from previous treatment must have elapsed prior to registration, with evidence for disease progression as outlined in inclusion criteria #2.
6. Age ≥18 years.
7. Life expectancy of greater than 12 weeks.
8. Eastern Cooperative Oncology Group [ECOG] performance status of 2 or less
9. Pts must have near normal organ and marrow function within 2 weeks prior to registration as defined below:

   * Granulocytes > 1500/mm³
   * Platelet count > 100,000/mm³
   * Bilirubin < 1.5 mg/dL
   * Serum glutamate pyruvate transaminase (ALT) < 2 times the institutional upper limit of normal
   * Creatinine < 1.5 mg/dL or a calculated creatinine clearance > 50 mL/min
10. Pts with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for 5 years or more (excluding non-melanomatous skin cancers treated with curative intent).
11. All sites of disease must be evaluated within 4 weeks prior to registration.
12. Have the ability to understand the requirements of the study, provide written informed consent and authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

1. The use of bisphosphonates (i.e. pamidronate sodium or zoledronic acid) will be allowed provided that the patient has been receiving that medication for 4 weeks or more with evidence of progressive disease as outlined above.

   • Pts will not be allowed to start bisphosphonate while receiving protocol treatment unless clinically indicated (will need approval of the study principal investigator). Those patients already on a bisphosphonate will need to continue to receive the bisphosphonate as previously scheduled.
2. Pts must not have had prior radiotherapy within 4 weeks prior to registration. Patient cannot have had prior Strontium 89, Samarium 153, or other radioisotope.

   • If a pt requires palliative radiotherapy, two consecutive rises (baseline value must be obtained after completion of radiation treatment) in PSA measurement are necessary, each separated from the previous by a minimum of two weeks.
3. No concurrent use of estrogen, or estrogen-like agents (i.e. PC-SPES, Saw Palmetto, or other herbal products which may contain phytoestrogens), or any other hormonal therapy (including megastrol acetate, finasteride, ketoconazole, and systemic corticosteroids) is allowed at any time during the study. Prior use of these agents will need to be discontinued 4 weeks or more prior to enrollment. Disease progression needs to be confirmed as outlined in inclusion criteria #2.
4. Pts with type I insulin-dependent diabetes or poorly-controlled type II insulin-dependent diabetes or a fasting blood glucose of more than 10 mmol/L (200 mg/dL) will be excluded due to difficulty evaluating the tumor metabolic activity using FDG-PET.
5. Patients must not have active angina pectoris, or known heart disease of New York Heart Association Class III-IV. Patients must not have a history of myocardial infarction within 6 months prior to registration. No history or evidence of ventricular dysrhythmias or other unstable arrythmia is allowed (rate controlled atrial fibrillation is allowed if the patient is asymptomatic from a cardiac standpoint).
6. Patients must not have any known history of carcinomatous meningitis or brain metastases.
7. No serious concurrent medical illness or active infection should be present which would jeopardize the ability of the patient to receive the therapy outlined in this protocol with reasonable safety.
8. No major surgery within 21 days of starting treatment with Panzem NCD.
9. Pts must not receive any investigational agents other than Panzem NCD for the duration of their participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
6 month progression free survival | at time of progression

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Derived] Harrison MR, Hahn NM, Pili R, Oh WK, Hammers H, Sweeney C, Kim K, Perlman S, Arnott J, Sidor C, Wilding G, Liu G. A phase II study of 2-methoxyestradiol (2ME2) NanoCrystal(R) dispersion (NCD) in patients with taxane-refractory, metastatic castrate-resistant prostate cancer (CRPC). Invest New Drugs. 2011 Dec;29(6):1465-74. doi: 10.1007/s10637-010-9455-x. Epub 2010 May 25. PMID 20499131